CLINICAL TRIAL: NCT02601820
Title: The Patient-Reported Outcomes Project of HCV-TARGET (PROP UP)
Brief Title: The Patient-Reported Outcomes Project of HCV-TARGET
Acronym: PROP-UP
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1633
Record Dates: First submitted 2015-11-03; First posted 2015-11-10 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C, Chronic; Liver Diseases
Keywords: patient-reported outcomes; observational; HCV; Hepatitis C; Liver Disease; Liver; Infectious Disease; PROs
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Hepatitis C; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The PROP UP research study is funded by The Patient Centered Outcomes Research Institute (PCORI). PROP UP is a multi-centered prospective observational study that will evaluate all-oral treatment regimens for chronic hepatitis C viral (HCV) infection regarding several patient-reported outcomes (PROs) such as HCV-associated symptoms, treatment side effects, medication adherence, out of pocket costs, comorbid conditions, and long-term benefits of cure and harms of treatment to compare PROs of different treatment regimens, treatment durations, and patient subgroups. Participants will be recruited from 9 U.S. liver centers. Approximately 1920 patients with HCV infection who are prescribed a regimen containing Sofosbuvir/Ledipasvir(SOF/LED), SOF/Velpatasvir(SOF/VEL), Grazoprevir/Elbasvir(GRZ/ELB), OBV/PTV/r + DSV (PRoD), or daclatasvir/SOF (DAC/SOF) will be recruited and approximately 1600 patients who are approved and begin HCV treatment will be enrolled in the longitudinal study. PRO surveys will be evaluated before, during and after HCV treatment.

PROP UP is a collaborative effort between behavioral and biomedical researchers, a patient engagement group and a patient advocacy organization.

DETAILED DESCRIPTION:
Newer, more effective all-oral regimens for hepatitis C viral (HCV) infection are available. However the available data from industry-sponsored trials do not provide all the information that patients need, nor do these data represent the broad spectrum of patients treated in real-world practice. Trials also exclude disadvantaged subgroups, focus on short-term efficacy and clinician-rated adverse events, rarely obtain the patient's perspective, and do not investigate longer-term harms of treatment or benefits of viral cure. Given these informational gaps, patient-centered outcomes research on treatment harms and benefits that matter most to patients, is needed.

PROP UP is funded by The Patient Centered Outcomes Research Institute (PCORI). PROP UP is a multi-centered prospective observational study that will evaluate newly approved direct acting antiviral (DAA) treatment regimens for HCV regarding several patient-reported outcomes (PROs) such as HCV-associated symptoms, treatment side effects, medication adherence, out of pocket costs, comorbid conditions, and long-term benefits of cure and harms of treatment to compare PROs of different treatment regimens, treatment durations, and patient subgroups.

PROP UP is a collaborative effort between researchers, a patient engagement group, and a patient advocacy organization. Eleven U.S. liver centers will collaborate on PROP UP. Approximately 1920 patients with HCV infection who are prescribed a DAA regimen for chronic HCV will be consented and will complete baseline PRO surveys. Approximately 1600 patients who are approved and begin HCV treatment will be enrolled in the longitudinal study. Participants will complete several PRO surveys at 5 assessment periods during the study: baseline, treatment week 4, end of treatment, 3 months post-treatment, and 12 months post-treatment. PRO survey data will be collected via 3 options: patient home-based computers, tablet, smartphone; phone-administered surveys with a centralized call enter; or at regular clinic visits.

Analysis of PROs collected longitudinally before, during and after treatment for HCV will allow the investigators to answer a variety of questions important to patients and clinicians. Specifically, the investigators will evaluate: (a) prevalence of pre-existing baseline symptoms associated with HCV; (b) the development of new onset treatment side effects and exacerbation of pre-existing symptoms during HCV treatment; (c) medication adherence and out of pocket costs associated with treatment; (d) changes in HCV-associated symptoms and functional status in patients who are cured; (e) long-term patient-reported harms associated with treatments and long-term benefits associated with viral cure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCV genotype 1-6
* English-speaking
* Age 21 or older
* Medically cleared and being prescribed one of the following DAA regimens:

  * sofosbuvir/ledipasvir (SOF/LED) with or without ribavirin
  * ombitasvir/paritaprevir/ritonavir with dasabuvir (PRoD), with or without ribavirin
  * elbasvir/grazoprevir (ELB/GRZ) with or without ribavirin
  * daclatasvir/sofosbuvir, with or without ribavirin (DAC/SOF)
  * sofosbuvir/velpatasvir (SOF/VEL)

Exclusion Criteria:

* Inability to provide written informed consent
* Currently participating in a pharmaceutical-sponsored drug trial of hepatitis C treatment
* Major cognitive or mental impairment
* Unable to read or speak English
* Unwilling or unable to complete survey questionnaires

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated for Hep C treatment in 9 large academic liver centers and two private gastroenterology practices in the US.
Sampling Method: Non-Probability Sample
Enrollment: 1601 (Actual)
Dates: Start 2015-11; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna M. Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (11):
- United States (11):
  - University of California at Davis, Davis, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Rush University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - St Louis University, St Louis, Missouri
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serper M, Evon DM, Amador J, Stewart PW, Sarkar S, Lok AS, Sterling RK, Reeve BB, Golin CE, Rajender Reddy K, Lim JK, Reau N, Nelson DR, Di Bisceglie AM, Fried MW. Patient-reported outcomes 12 months after hepatitis C treatment with direct-acting antivirals: Results from the PROP UP study. Liver Int. 2021 Apr;41(4):692-704. doi: 10.1111/liv.14781. Epub 2021 Jan 22. PMID 33387381
- [Derived] Evon DM, Sarkar S, Amador J, Lok AS, Sterling RK, Stewart PW, Reeve BB, Serper M, Reau N, Rajender Reddy K, Di Bisceglie AM, Nelson DR, Golin CE, Lim JK, Fried MW. Patient-reported symptoms during and after direct-acting antiviral therapies for chronic hepatitis C: The PROP UP study. J Hepatol. 2019 Sep;71(3):486-497. doi: 10.1016/j.jhep.2019.04.016. Epub 2019 May 13. PMID 31096006
- [Derived] Evon DM, Stewart PW, Amador J, Serper M, Lok AS, Sterling RK, Sarkar S, Golin CE, Reeve BB, Nelson DR, Reau N, Lim JK, Reddy KR, Di Bisceglie AM, Fried MW. A comprehensive assessment of patient reported symptom burden, medical comorbidities, and functional well being in patients initiating direct acting antiviral therapy for chronic hepatitis C: Results from a large US multi-center observational study. PLoS One. 2018 Aug 1;13(8):e0196908. doi: 10.1371/journal.pone.0196908. eCollection 2018. PMID 30067745
- [Derived] Evon DM, Golin CE, Stewart P, Fried MW, Alston S, Reeve B, Lok AS, Sterling RK, Lim JK, Reau N, Sarkar S, Nelson DR, Reddy KR, Di Bisceglie AM. Patient engagement and study design of PROP UP: A multi-site patient-centered prospective observational study of patients undergoing hepatitis C treatment. Contemp Clin Trials. 2017 Jun;57:58-68. doi: 10.1016/j.cct.2017.03.013. Epub 2017 Mar 22. PMID 28342989
- See also: PROP UP Patient Website — http://propup.web.unc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 liver or gastroenterology centers in the United States: 9 academic medical centers, 2 private gastroenterology centers.
  1601 patients officially enrolled who provided informed consent, completed baseline patient-reported outcome (PRO) surveys and were prescribed one of five direct acting antiviral treatment regimens for chronic hepatitis C.
Pre-assignment Details: None. Observational study included enrolled patients who completed PRO data at follow-up time periods.
Groups:
- Chronic HCV Patients During and After HCV Treatment: 1601 patients with chronic hepatitis C were enrolled. Criteria for enrollment included: providing consent, completing baseline patient-reported outcome (PRO) measures, and initiating one of five direct acting antiviral (DAAs) therapy.
Period: Pre-Treatment (T1)
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Started | 1601 (1601 patients were enrolled and completed Baseline PROs (T1).)
Completed | 1601
Not Completed | 0
Period: Early On-Treatment (T2)
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Started | 1584 (Of 1601, 17 were excluded at T2 due to death, withdrawal, other reason. 1584 remained in the study.)
Completed | 1533 (Of 1584, 51 were excluded for a missing T2 record. 1533 provided data at T2. Some outcomes missing.)
Not Completed | 51
Not completed — Missing T2 Record | 51
Period: Late On-Treatment (T3)
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Started | 1573 (Of 1601, 28 were excluded at T3 due to death, withdrawal, other reason. 1573 remained in the study.)
Completed | 1524 (Of 1573, 49 were excluded for a missing T3 record. 1524 provided data at T3. Some outcomes missing.)
Not Completed | 49
Not completed — missing T3 Record | 49
Period: 12 Weeks Post-Treatment (T4)
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Started | 1564 (Of 1601, 37 were excluded at T4 due to death, withdrawal, other reason. 1564 remained in the study.)
Completed | 1561 (Of 1564, 3 were excluded for a missing T4 record. 1561 provided data at T4. Some outcomes missing.)
Not Completed | 3
Not completed — Missing T4 record | 3
Period: 1-Yr Post-Treatment (T5)
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Started | 1528 (Of 1601, 73 were excluded at T5 due to death, withdrawal, other reason. 1528 remained in the study.)
Completed | 1440 (Of 1528, 88 were excluded for a missing T5 record. 1440 provided data at T5. Some outcomes missing.)
Not Completed | 88
Not completed — Missing T5 Record | 88

BASELINE CHARACTERISTICS:
Groups:
- Chronic HCV Patients on Treatment: All 1,601 patients with chronic HCV enrolled at baseline
Arm/Group | Chronic HCV Patients on Treatment
Number analyzed (Participants) | 1601
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 714
  Male | 887
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66
  Not Hispanic or Latino | 1260
  Unknown or Not Reported | 275
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 519
  White | 975
  More than one race | 32
  Unknown or Not Reported | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1601
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Depression-8 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Depression-8a range from 38.2 - 81.3. Higher scores indicate worse symptoms. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points.Higher scores indicate worse Depression. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1598
    (all) | 49.3 (10.5)
PROMIS Anger [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Anger-5 item short form at baseline (T1) prior to starting HCV Treatment. Higher scores indicate worse Anger/irritability.
  PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Anger-5a range from 32.9 - 82.9. Higher scores indicate worse symptoms. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points.
  units on a scale | 48.9 (11.2)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Anxiety-4 item short form at baseline (T1) prior to starting HCV Treatment.
  PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Anxiety-4a range from 40.3 - 81.6. Higher scores indicate worse symptoms. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points.
  Higher scores indicate worse Anxiety. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1591
    (all) | 50.4 (10.2)
PROMIS Cognitive Concerns [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Applied Cognitive-General Concerns 8 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Applied Cognitive-General Concerns-8a range from 22.41 - 63.48. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points.Higher scores indicate worse Cognitive Concerns. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1599
    (all) | 33 (9.0)
PROMIS Pain Interference [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Pain Interference 8 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Pain Interference-8a range from 40.7 - 77.0. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points. Higher scores indicate worse Pain Interference. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1600
    (all) | 53 (11)
PROMIS Fatigue [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Fatigue-7a item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Fatigue 7a short form range from 29.4 -83.2. Higher scores indicate worse symptoms. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points.Higher scores indicate worse Fatigue. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1599
    (all) | 51.8 (10.8)
PROMIS Sleep Disturbance [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Sleep Disturbance-8a short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Sleep Disturbance-8a short form scores range from 28.9 - 76.5. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points. Higher scores indicate worse Sleep Disturbance. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1600
    (all) | 51.8 (11.4)
PROMIS Abdominal Pain [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Belly Pain-5 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Belly Pain-5a range from 39.3 - 80. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points. Higher scores indicate worse Belly Pain. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1600
    (all) | 36.1 (12.9)
PROMIS Diarrhea [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Diarrhea-6 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Diarrhea-6a range from 45.9 - 75.2. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points. Higher scores indicate worse Diarrhea. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1584
    (all) | 35.6 (8.7)
PROMIS Nausea and Vomiting [Mean (Standard Deviation); unit: units on a scale] — Patients completed the PROMIS Nausea and Vomiting-4 item short form at baseline (T1) prior to starting HCV Treatment. PROMIS raw scores are converted to standardized T-scores, with a mean of 50 and standard deviation of 10. T-scores for the PROMIS Nausea and Vomiting 4a scale range from 45.0 - 80.1. Studies in other medical populations suggest that the minimally important difference generally ranges from 2-5 points. Higher scores indicate worse Nausea/Vomit. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1585
    (all) | 41.6 (8.5)
Headache Impact Test (HIT-6) [Mean (Standard Deviation); unit: units on a scale] — Patients completed the Headache Inventory Test-6 at baseline (T1) prior to starting HCV Treatment. The six items are scored on a 5-point likert scale ranging from never to always. The final score is summed and can range from 36-78, with higher scores indicate worse headaches. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1577
    (all) | 45.3 (10)
TMSAS Overall Symptom Burden [Mean (Standard Deviation); unit: units on a scale] — Overall symptom burden was measured using the Memorial Symptom Assessment Scale (MSAS). The MSAS is a reliable and validated 32-item instrument used to measure change in pre-existing HCV symptoms. The MSAS evaluates 32 symptoms common in medical populations. Patients indicate the presence or absence of a symptom. If present, rate the construct on severity, frequency and distress. An overall symptom burden score is created: TMSAS (total MSAS score). The TMSAS scores range from 0 (no symptom) to 4 (present, severe, frequent, distressing). Higher scores indicate worse overall symptom burden. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1589
    (all) | 0.6 (0.5)
HCV-PRO Functional Well-Being [Mean (Standard Deviation); unit: units on a scale] — Patients completed the HCV-PRO at baseline (T1) prior to starting HCV Treatment. The HCV-PRO is new disease specific measure. It has 16 items with responses ranging from 1-5 with the sum transformed to a 0-100 scale. Higher scores indicate better functional well-being. Population: 1601 patients were enrolled and have a PRO Completion Record. Lower numbers in each PRO row below due to missing data.
  units on a scale
    number analyzed (Participants) | 1493
    (all) | 71.7 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Memorial Symptom Assessment Scale Mean Score (TMSAS) From Baseline to On-Treatment
Description: Change in "Overall Symptom Burden" was measured using the Memorial Symptom Assessment Scale (MSAS). Patients indicate the presence or absence of a symptom, and if present, rate the symptom on severity, frequency and interference. The total MSAS score (TMSAS) can range from 0 (no symptom) to 4 (symptom present and worst severity, frequency and distress). Change in TMSAS score is calculated as Baseline TMSAS mean score minus T2 TMSAS mean score or Baseline TMSAS mean score minus T3 TMSAS mean score.
  Change scores could range from +/- 4.0. Higher scores (+) indicate worse symptom burden.
  To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in the TMSAS = 0.3 points; therefore TMSAS change scores > +/- 0.3 were considered clinically meaningful.
Time Frame: Baseline to up to 24 weeks of HCV Treatment
Population: Of 1533 patients with complete record at T2, 1517 provided sufficient TMSAS data to calculate change score.
  Of 1524 patients with complete record at T3, 1513 provided sufficient TMSAS data to calculate change score.
  Discrepancies due to missing TMSAS data at T2 or T3.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients on Therapy: All enrolled patients with MSAS data available at T2 or T3 during HCV treatment
Arm/Group | Chronic HCV Patients on Therapy
Number analyzed (Participants) | 1533
units on a scale
  Change in TMSAS score from T1 to T2 | -0.10 [-0.10 to -0.10]
  Change in TMSAS score from T1 to T3: number analyzed (Participants) | 1524
  Change in TMSAS score from T1 to T3 | -0.1 [-0.10 to -0.10]

2. Secondary Outcome: Change in Treatment-Related Symptom Mean Scores From Baseline to On-Treatment
Description: Change in Treatment-Related Symptoms was measured using multiple surveys from the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) and the Headache Impact Test (HIT-6). Mean CHANGE Scores were calculated as baseline mean score minus T2 mean score or baseline mean score minus T3 mean score. Lower change scores (-) indicate symptoms improved.
  1. PROMIS Fatigue-7 mean change score range = +/- 53.9
  2. PROMIS Sleep Disturbance-8a mean change score range = +/- 47.1
  3. PROMIS Nausea/Vomiting-4 mean change score range = +/- 44.0
  4. PROMIS Diarrhea-6 mean change score range = +/- 42.8
  5. PROMIS Anger-5 mean change score range = +/- 50.5.
  6. PROMIS Anxiety-4 mean change score range = +/- 41.4
  7. HIT-6 mean change score range = +/- 42
  To aid in interpretation of clinical significance, a 5% change from baseline is considered a "minimally important change (MIC)." The 5% MIC change in a PROMIS or HIT-6 score is +/- 2.5 points.
Time Frame: Baseline to up to 24 weeks of HCV Treatment
Population: Sample size may differ for each mean change score due to missing survey data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients on Therapy: All enrolled patients with symptom data recorded at T2 or T3 during HCV treatment
Arm/Group | Chronic HCV Patients on Therapy
Number analyzed (Participants) | 1533
units on a scale
  Change in Fatigue Mean Score from T1 to T2: number analyzed (Participants) | 1527
  Change in Fatigue Mean Score from T1 to T2 | -1.1 [-1.6 to -0.6]
  Change in Sleep disturbance score from T1 to T2: number analyzed (Participants) | 1526
  Change in Sleep disturbance score from T1 to T2 | -1.6 [-2.1 to -1.1]
  Change in Nausea/Vomiting mean score from T1 to T2: number analyzed (Participants) | 1499
  Change in Nausea/Vomiting mean score from T1 to T2 | 0.8 [0.3 to 1.2]
  Change in Diarrhea mean score from T1 to T2: number analyzed (Participants) | 1498
  Change in Diarrhea mean score from T1 to T2 | 0.8 [0.4 to 1.3]
  Change in Irritability mean score from T1 to T2: number analyzed (Participants) | 1525
  Change in Irritability mean score from T1 to T2 | -1.2 [-1.8 to -0.7]
  Change in Anxiety mean score from T1 to T2: number analyzed (Participants) | 1496
  Change in Anxiety mean score from T1 to T2 | -1.5 [-2.0 to -1.1]
  Change in headache HIT-6 mean score from T1 to T2: number analyzed (Participants) | 1490
  Change in headache HIT-6 mean score from T1 to T2 | 0.2 [-0.3 to 0.6]
  Change in Fatigue mean score from T1 to T3: number analyzed (Participants) | 1519
  Change in Fatigue mean score from T1 to T3 | -1.1 [-1.6 to -0.6]
  Change in sleep disturbance score from T1 to T3: number analyzed (Participants) | 1522
  Change in sleep disturbance score from T1 to T3 | -1.8 [-2.3 to -1.3]
  Change in nausea/vomiting mean score from T1 to T3: number analyzed (Participants) | 1496
  Change in nausea/vomiting mean score from T1 to T3 | -0.2 [-0.6 to 0.3]
  Change in Diarrhea mean score from T1 to T3: number analyzed (Participants) | 1500
  Change in Diarrhea mean score from T1 to T3 | 0.6 [0.1 to 1.1]
  Change in anger mean score from T1 to T3: number analyzed (Participants) | 1522
  Change in anger mean score from T1 to T3 | -0.8 [-1.3 to -0.2]
  Change in anxiety mean score from T1 to T3: number analyzed (Participants) | 1499
  Change in anxiety mean score from T1 to T3 | -1.4 [-1.9 to -0.9]
  Change in headache HIT-6 mean score from T1 to T3: number analyzed (Participants) | 1479
  Change in headache HIT-6 mean score from T1 to T3 | -0.1 [-0.5 to 0.4]

3. Secondary Outcome: Change in HCV-PRO Mean Scores From Baseline to On-Treatment
Description: HCV-specific Functional Well-Being was measured using the disease-specific "HCV-PRO." The scale includes 16 items that measure physical, emotional and social functioning, productivity, intimacy, and perception of quality of life.
  The Means provided are the HCV-PRO Mean Change Scores, calculated as Baseline HCV-PRO mean score minus T2 HCV-PRO mean score or Baseline HCV-PRO mean score minus T3 HCV-PRO mean score.
  HCV-PRO mean change scores range from +/- 100. Higher change scores (+) indicate better HCV-PRO outcomes.
  To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in HCV-PRO = 4 points; therefore HCV-PRO change scores > +/- 4.0 were considered clinically meaningful.
Time Frame: Baseline to up to 24 weeks of HCV Treatment
Population: Of 1533 patients with data records at T2, 1346 had analyzable HCV-PRO data at T2.
  Of 1524 patients with data records at T3, 1356 had analyzable HCV-PRO data at T3. Discrepancies due to missing HCV-PRO data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients on Therapy: All enrolled patients with HCV-PRO data available at T2 or T3 during HCV treatment
Arm/Group | Chronic HCV Patients on Therapy
Number analyzed (Participants) | 1533
units on a scale
  Change in HCV-PRO mean score from T1 to T2: number analyzed (Participants) | 1346
  Change in HCV-PRO mean score from T1 to T2 | 3.2 [2.3 to 4.0]
  Change in HCV-PRO mean score from T1 to T3: number analyzed (Participants) | 1356
  Change in HCV-PRO mean score from T1 to T3 | 3.8 [2.8 to 4.7]

4. Secondary Outcome: Cumulative Out of Pocket Costs During HCV Treatment
Description: Cumulative out of pocket (OOP) costs incurred by patients during HCV treatment was measured by a survey recording 5 direct and 5 indirect costs of treatment. OOP costs were collected early on-treatment (T2), late on-treatment (T3), and early post-treatment (T4) in case patients paid bills after treatment ended.
  The Mean is the average dollar ($$) amount for Total OOP Cost of HCV Treatment for the cohort, calculated by summing the OOP costs for each patient reported at T2+T3+T4.
Time Frame: Up to 24 weeks of HCV Treatment
Population: Of 1601 patients enrolled, OOP cost data was recorded by 1578 patients. Due to unreliable data, especially at the upper limit, 40 cases (2.53%) were eliminated from each tail (lower and upper limit), totaling 80 cases (5.06%) of the 1578 sample. OOP dollar amount below based on 1498 cases.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients During and After HCV Treatment: 1601 patients with chronic HCV were enrolled. Criteria for enrollment included: providing consent, completing baseline patient-reported outcome (PRO) measures, and initiating one of five direct acting antiviral (DAAs) therapy.
Arm/Group | Chronic HCV Patients During and After HCV Treatment
Number analyzed (Participants) | 1498
units on a scale | 582.50 [490.60 to 674.30]

5. Secondary Outcome: Percentage of Participants With Nonadherence During HCV Treatment
Description: Medication adherence was measured using the Voils' Medication Adherence Survey (VMAS). The VMAS consists of 3 items that evaluated the extent of adherence using a 5-point Likert scale from 1=None of the time to 5=All of the time. The 3 items assess how often participants missed doses, skip doses, or do not take doses over the past 7 days and are averaged into a single score. A dichotomous variable was created to categorize patients as 100% (adherent) or <100% (nonadherent) during HCV treatment at early treatment (T2) and late treatment (T3).
Time Frame: Up to 24 weeks of HCV Treatment
Population: Of 1601 enrolled patients, 1562 had VMAS adherence data at either early treatment (T2) or late treatment (T3). 1513 patients had adherence data at T2. 1476 patients had adherence data at T3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Patients With Baseline Mental Health Disturbance; Patients Without Baseline Mental Health Disturbance: For this analysis, participants were classified as having mental health disturbances if they reported taking psychiatric medications for psychiatric conditions at enrollment or had ever been hospitalized for a psychiatric condition.
- Patients With Baseline Alcohol Abuse; Patients Without Baseline Alcohol Abuse: for this analysis, current alcohol abuse was evaluated using a score of greater than or equal to 5 on the Substance Abuse Mental Illness Symptom Screener (SAMISS), using questions similar to the Alcohol Use Disorders Identification Test (AUDIT).
- Patients With Baseline Substance Use; Patients Without Baseline Substance Use: For this analysis, substance abuse was classified as self-reported use of prescription drugs to either get high or change the way a patient feels, or use of nonprescription street drugs within the year prior to enrollment using the SAMISS screener.
Arm/Group | Patients With Baseline Mental Health Disturbance | Patients Without Baseline Mental Health Disturbance | Patients With Baseline Alcohol Abuse | Patients Without Baseline Alcohol Abuse | Patients With Baseline Substance Use | Patients Without Baseline Substance Use
Number analyzed (Participants) | 1562 | 1562 | 1562 | 1562 | 1562 | 1562
percentage of participants
  Nonadherence rate (%) early on-treatment (T2): number analyzed (Participants) | 550 | 957 | 221 | 1285 | 344 | 1163
  Nonadherence rate (%) early on-treatment (T2) | 4.5 [3.1 to 6.6] | 4.2 [3.1 to 5.6] | 5.9 [3.5 to 9.8] | 4 [3.1 to 5.3] | 5.5 [3.6 to 8.5] | 4.3 [3.0 to 5.2]
  Nonadherence rate (%) late on-treatment (T3): number analyzed (Participants) | 546 | 924 | 212 | 1257 | 332 | 1137
  Nonadherence rate (%) late on-treatment (T3) | 9 [6.9 to 11.7] | 7.6 [6.0 to 9.5] | 13.7 [9.7 to 19.0] | 7.2 [5.9 to 8.7] | 9 [6.4 to 12.6] | 7.8 [6.4 to 9.5]

6. Secondary Outcome: Change in Total Memorial Symptom Assessment Scale (TMSAS) Mean Score From Baseline to 3-months Post Treatment
Description: Change in "Overall Symptom Burden" from Baseline to 3-months post-treatment was measured using the Memorial Symptom Assessment Scale (MSAS).
  The total Overall Symptom Burden mean change score (TMSAS) was calculated as Baseline TMSAS mean score minus T4 TMSAS mean score.
  Lower scores (-) indicate better outcomes. Change scores were calculated for two subgroups: (1) Patients who achieved SVR and (2) patients who did not achieve SVR.
  TMSAS Mean Change Scores could range from +/- 4.
  To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in the TMSAS = 0.3 points; therefore TMSAS change scores > +/- 0.3 were considered clinically meaningful.
Time Frame: Baseline to 3-months post-treatment
Population: Of 1601 patients enrolled, 1430 patients had post-treatment HCV RNA available to determine SVR status. Of these, 1362 achieved SVR, 68 did not achieve SVR. SVR data were missing on 171 patients. Additional missing numbers (from 1362 to 1313 and 68 to 58) were due to missing MSAS survey data at 3-months post-treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients Who Achieved SVR: Chronic HCV patients who achieved a sustained virologic cure (SVR) 3-months post-treatment
- Chronic HCV Patients Who Did Not Achieve SVR: Chronic HCV patients who did not achieve a sustained virologic cure (SVR) 3-months post-treatment
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1313 | 58
units on a scale | -0.2 [-0.2 to -0.2] | -0.1 [-0.2 to 0.0]

7. Secondary Outcome: Change in HCV Symptom Mean Scores From Baseline to 3-months Post Treatment
Description: Change in Symptoms was measured using surveys below. Change scores were calculated as baseline mean minus T4 mean. Lower change scores (-) indicate symptom improved
  1. PROMIS Fatigue mean change score range = +/- 53.9
  2. PROMIS Sleep Disturbance mean change score range = +/- 47.1
  3. PROMIS Nausea mean change score range = +/- 44.0
  4. PROMIS Diarrhea mean change score range = +/- 42.8
  5. PROMIS Anger mean change score range = +/- 50.5.
  6. PROMIS Anxiety mean change score range = +/- 41.4
  7. PROMIS Depression mean change score range = +/- 43.1
  8. PROMIS Cognitive Concern mean change score range = +/- 39.5
  9. PROMIS Pain mean change score range = +/- 36.4
  10. PROMIS Belly Pain mean change score range = +/- 50.2
  11. Headache HIT-6 mean change score range = +/- 42 A 5% change from baseline is considered the clinically "minimally important change" (MIC). The 5% MIC = +/- 2.5 points.
  Change scores were calculated for two subgroups: Patients who did and did not achieve SVR
Time Frame: Baseline to 3-months post-treatment
Population: Of 1601 patients enrolled, 1430 patients had post-treatment HCV RNA available to determine SVR status. Of these, 1362 achieved SVR, 68 did not achieve SVR. SVR data were missing on 171 patients. Missing numbers below are due to missing PRO survey data at T4.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1362 | 68
units on a scale
  Depression change score: number analyzed (Participants) | 1326 | 59
  Depression change score | -2.3 [-2.8 to -1.8] | 0.2 [-1.7 to 2.1]
  Anger change score: number analyzed (Participants) | 1327 | 59
  Anger change score | -2.1 [-2.7 to -1.5] | 0.7 [-1.9 to 3.4]
  Anxiety change score: number analyzed (Participants) | 1310 | 58
  Anxiety change score | -1.7 [-2.2 to -1.2] | -0.7 [-3.0 to 1.5]
  Cognitive Concerns change score: number analyzed (Participants) | 1326 | 59
  Cognitive Concerns change score | -1.4 [-1.8 to -0.9] | 0 [-1.7 to 1.8]
  Pain Interference change score: number analyzed (Participants) | 1327 | 59
  Pain Interference change score | -2.3 [-2.8 to -1.8] | -1.7 [-4.1 to 0.7]
  Fatigue change score: number analyzed (Participants) | 1329 | 58
  Fatigue change score | -4.1 [-4.6 to -3.5] | -2.9 [-5.4 to -0.4]
  Sleep change score: number analyzed (Participants) | 1327 | 59
  Sleep change score | -3.1 [-3.6 to -2.5] | -0.9 [-3.3 to 1.4]
  Belly Pain change score: number analyzed (Participants) | 1326 | 58
  Belly Pain change score | -2.3 [-2.9 to -1.6] | 0.9 [-1.9 to 3.6]
  Diarrhea change score: number analyzed (Participants) | 1308 | 58
  Diarrhea change score | -0.1 [-0.6 to 0.4] | 0.7 [-2.1 to 3.5]
  Nausea change score: number analyzed (Participants) | 1308 | 59
  Nausea change score | -1.5 [-1.9 to -1.0] | -0.3 [-2.1 to 1.6]
  Headache change score: number analyzed (Participants) | 1297 | 55
  Headache change score | -1.5 [-1.9 to -1.0] | -1.1 [-3.1 to 0.9]

8. Secondary Outcome: Change in HCV-PRO Mean Score From Baseline to 3-months Post Treatment
Description: HCV-specific Functional Well-Being was measured using the disease-specific "HCV-PRO."
  The means provided are the HCV-PRO Mean Change Scores, calculated as Baseline HCV-PRO mean score minus T4 HCV-PRO mean score. Change scores were calculated for two subgroups: (1) Patients who achieved SVR and (2) patients who did not achieve SVR.
  HCV-PRO Mean Change Scores could range from +/- 100. Higher change scores (+) indicate better HCV-PRO outcomes.
  To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in HCV-PRO = 4 points; therefore HCV-PRO change scores > +/- 4.0 were considered clinically meaningful.
Time Frame: Baseline to 3-months post-treatment
Population: Of 1601 patients enrolled, 1430 patients had post-treatment HCV RNA available to determine SVR status. Of these, 1362 achieved SVR, 68 did not achieve SVR. SVR data were missing on 171 patients. Additional missing numbers due to missing HCV-PRO survey data at 3-months post-treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1172 | 54
units on a scale | 6.5 [5.5 to 7.5] | 2.0 [-7.1 to 3.1]

9. Secondary Outcome: Change in Total Memorial Symptom Assessment Scale (TMSAS) Mean Score From Baseline to 1 Year Post-Treatment
Description: Change in "Overall Symptom Burden" from Baseline to 1 year post-treatment was measured using the Memorial Symptom Assessment Scale (MSAS). The total Overall Symptom Burden mean change score (TMSAS) was calculated as Baseline TMSAS mean score minus T5 TMSAS mean score.
  Lower scores (-) indicate better outcomes. Change scores were calculated for two subgroups: (1) Patients who achieved SVR and (2) patients who did not achieve SVR.
  TMSAS Mean Change Scores could range from +/- 4. To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in the TMSAS = 0.3 points; therefore TMSAS change scores > +/- 0.3 were considered clinically meaningful
Time Frame: Baseline to 1 year post-treatment
Population: 1430 of 1601 patients had post-treatment HCV RNA available to determine SVR status: 1362 achieved SVR, 68 did not. SVR data were missing on 171 patients. Of 1430, T5 records were missing for 93 cases (1337 remaining). Of the remaining 1337 records, TMSAS data were missing for 17 patients (1320 remaining: 1269 with SVR, 51 with no SVR)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Chronic HCV Patients Who Achieved SVR: Chronic HCV patients who achieved a sustained virologic cure (SVR) and completed PRO data one-year post-treatment (T5)
- Chronic HCV Patients Who Did Not Achieve SVR: Chronic HCV patients who did not achieve a sustained virologic cure (SVR) and completed data one-year post-treatment (T5)
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1269 | 51
units on a scale | -0.2 [-0.2 to -0.1] | 0 [-0.2 to 0.1]

10. Secondary Outcome: Changes in HCV Symptom Mean Scores From Baseline to 1 Year Post-Treatment
Description: Change in Symptoms was measured using surveys below. Change scores were calculated as baseline mean minus T5 mean. Lower change scores (-) indicate symptom improved
  1. PROMIS Fatigue mean change score range = +/- 53.9
  2. PROMIS Sleep Disturbance mean change score range = +/- 47.1
  3. PROMIS Nausea mean change score range = +/- 44.0
  4. PROMIS Diarrhea mean change score range = +/- 42.8
  5. PROMIS Anger mean change score range = +/- 50.5.
  6. PROMIS Anxiety mean change score range = +/- 41.4
  7. PROMIS Depression mean change score range = +/- 43.1
  8. PROMIS Cognitive Concern mean change score range = +/- 39.5
  9. PROMIS Pain mean change score range = +/- 36.4
  10. PROMIS Belly Pain mean change score range = +/- 50.2
  11. Headache HIT-6 mean change score range = +/- 42 A 5% change from baseline is considered the clinically "minimally important change" (MIC). The 5% MIC = +/- 2.5 points.
  Change scores were calculated for two subgroups: Patients who did and did not achieve SVR
Time Frame: Baseline to 1 year post-treatment
Population: 1430 patients had post-treatment HCV RNA available to determine SVR status: 1362 achieved SVR, 68 did not. SVR data were missing on 171 patients. T5 records were missing for 93 cases. Discrepancies from 1362 and 68 due to missing survey data at T5 for specific measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1285 | 52
units on a scale
  Depression change score: number analyzed (Participants) | 1277 | 52
  Depression change score | -2.2 [-2.7 to -1.7] | -0.9 [-2.8 to 1.0]
  Anger change score: number analyzed (Participants) | 1276 | 52
  Anger change score | -2.2 [-2.8 to -1.6] | -0.3 [-3.2 to 2.6]
  Anxiety change score: number analyzed (Participants) | 1264 | 51
  Anxiety change score | -2.0 [-2.5 to -1.4] | -0.4 [-2.3 to 1.6]
  Cognitive Concern change score: number analyzed (Participants) | 1277 | 52
  Cognitive Concern change score | -1.7 [-2.1 to -1.3] | 0.3 [-1.7 to 2.3]
  Pain Interference change score: number analyzed (Participants) | 1278 | 52
  Pain Interference change score | -1.9 [-2.5 to -1.4] | -0.8 [-3.4 to 1.9]
  Fatigue change score: number analyzed (Participants) | 1278 | 52
  Fatigue change score | -3.6 [-4.2 to -3.1] | -0.6 [-3.1 to 1.8]
  Sleep Disturbance change score: number analyzed (Participants) | 1278 | 52
  Sleep Disturbance change score | -3.1 [-3.7 to -2.5] | -1.3 [-4.2 to 1.6]
  Belly Pain change score: number analyzed (Participants) | 1276 | 52
  Belly Pain change score | -2.6 [-3.3 to -1.9] | -3.7 [-7.5 to 0.0]
  Diarrhea change score: number analyzed (Participants) | 1261 | 52
  Diarrhea change score | -0.3 [-0.8 to 0.2] | -0.1 [-2.8 to 2.6]
  Nausea change score: number analyzed (Participants) | 1260 | 52
  Nausea change score | -1.4 [-1.9 to -1.0] | -0.1 [-2.4 to 2.2]
  Headache HIT-6 Change score: number analyzed (Participants) | 1250 | 48
  Headache HIT-6 Change score | -1.5 [-2.0 to -1.1] | -0.7 [-2.2 to 0.9]

11. Secondary Outcome: Change in HCV-PRO Mean Score From Baseline to 1 Year Post-treatment
Description: HCV-specific Functional Well-Being was measured using the disease-specific "HCV-PRO." The scale includes 16 items that measure physical, emotional and social functioning, productivity, intimacy, and perception of quality of life.
  The Means provided are the HCV-PRO Mean Change Scores, calculated as Baseline HCV-PRO mean score minus T5 HCV-PRO mean score.
  Change scores were calculated for two subgroups: (1) Patients who achieved SVR and (2) patients who did not achieve SVR.
  HCV-PRO mean change scores could range from +/- 100. Higher change scores (+) indicate better HCV-PRO outcomes.
  To aid in interpretation of clinically significant change, a >5% change from baseline was set as the "minimally important change (MIC)" threshold. A 5% change in HCV-PRO = 4 points; therefore HCV-PRO change scores > +/- 4.0 were considered clinically meaningful.
Time Frame: Baseline to 1 year post-treatment
Population: 1430 of 1601 patients had post-treatment HCV RNA available to determine SVR status: 1362 achieved SVR, 68 did not. SVR data were missing on 171 patients. Of 1430, T5 records were missing for 93 cases (1337 remaining). Of the remaining 1337 records, HCV-PRO data were missing for 156 patients (1181 remaining: 1132 with SVR, 49 with no SVR)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chronic HCV Patients Who Achieved SVR | Chronic HCV Patients Who Did Not Achieve SVR
Number analyzed (Participants) | 1132 | 49
units on a scale | 7.0 [6.0 to 8.0] | 0.6 [-4.7 to 5.9]

ADVERSE EVENTS:
Time Frame: Up to 1.5 years from time of patient enrollment.
Description: This observational, non-interventional survey study did not systematically track NON-study related deaths, SAEs, or OAEs. Per protocol, only study-related deaths, SAEs, and OAEs were reportable and none occurred. All deaths observed were learned about inadvertently and via non-systematic methods during data collection processes. While possibly incomplete, the number reported represents all known observable deaths during the study. Other SAEs and OAEs were not monitored/assessed.
Arm/Group | Chronic HCV Patients During and After HCV Treatment
All-Cause Mortality (participants affected / at risk) | 34/1601
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The secondary outcome - cumulative out of pocket costs- may include less reliable data at the upper limit. Patient reporting of cumulative costs at 3 time points likely led to erroneous inflation affecting the upper limit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02601820/Prot_SAP_000.pdf